CLINICAL TRIAL: NCT00952718
Title: Effects of Inspiratory Muscle Training in Patients With Bronchiectasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Meng-Chih LIn, Vice Director, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CMRP-IRB-97-0458B
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Results first posted 2019-10-21 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Bronchiectasis
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): No intervention.
- Inspiratory muscle training (Experimental): With intervention.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — A pressure threshold device (Threshold® IMT HS730, RESPIRONICS Inc, Cedar Grove, NJ, USA) was used for the inspiratory muscle training program. The individualized training program was started at an intensity of 30% MIP, which was increased by 2 cmH2O each week, but the maximal intensity did not exceed 50% of MIP. Patients were encouraged to perform IMT for 30 minutes per day, at least 5 days a week for 8 weeks.
  Other Names: Pulmonary Rehabilitation
  Arms: Inspiratory muscle training

SUMMARY:
The purpose of this study is to determine whether inspiratory muscle training could improve and/or prevent the deterioration of inspiratory muscle strength, clinical cardiopulmonary outcome, systemic immunologic responses and quality of life in patients with bronchiectasis.

DETAILED DESCRIPTION:
Inspiratory muscle training is reportedly beneficial in patients with diverse chronic cardio-pulmonary diseases. It can increase inspiratory muscle strength and endurance, improves exercise capacity and quality of life (QOL), and decreases the perception of dyspnea (POD) for adults with stable chronic obstructive pulmonary disease (COPD). Though the pathophysiology in COPD and bronchiectasis are different, there are some similarities in clinical presentation. In COPD patients, lung hyperinflation induces functional weakness of the inspiratory muscle and increases elastic load to breathing and intrinsic positive end expiratory pressure. Patients with bronchiectasis shows reduced ratio of FEV1/FVC, reduced FEV1, and normal or slightly reduced FVC, which indicate that airways are blocked by mucus. However, there has been no study that used IMT as a training modality to determine its effect in bronchiectasis. The clinical relevance of increased respiratory muscle strength per se by IMT alone is unknown. This study tried to evaluate the feasibility and effectiveness of home-based threshold training and examined if the effects of IMT extends to clinical outcomes such as activities of daily living and QOL in bronchiectasis patients.

ELIGIBILITY:
Inclusion Criteria:

* Bronchiectasis confirmed by clinical history, pulmonary function test, and high resolution computed tomography

Exclusion Criteria:

* Had recent exacerbation within six weeks
* Use of corticosteroid
* With poor consciousness level
* Have cerebro-vascular or neuro-muscular disorders

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meng-Chih Lin, MD, Principal Investigator — Chang Gung Memorial Hospital-Kaohsiung Medical Center
Locations (1):
- Chang Gung Memorial Hospital-Kaohsiung Medical Center, Kaohsiung City, Taiwan

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Inspiratory Muscle Training
Started | 19 | 19
Completed | 13 | 13
Not Completed | 6 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inspiratory Muscle Training | Control | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (10) | 56 (9) | 60 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 6 | 7 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 13 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 13 | 13 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Maximum Inspiratory Pressure (MIP) and Maximum Expiratory Pressure (MEP) at 8 Weeks
Description: MEP was measured after maximal inspiration,while MIP was measured after maximal expiration with each subject seated and wearing a nose-clip. An experienced respiratory therapist strongly urged the subjects to make maximum inspiratory and expiratory efforts at or near residual and total lung capacity, respectively. Determinations were repeated until two technically satisfactory measurements were recorded, with the highest value used for calculations.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: cmH2O
Arm/Group | Inspiratory Muscle Training | Control
Number analyzed (Participants) | 13 | 13
cmH2O
  MIP baseline | 60 (21) | 71 (16.4)
  MIP at 8 weeks | 84 (29) | 69 (19)
  MEP at baseline | 72 (31) | 76 (20)
  MEP at 8 weeks | 104 (35) | 88 (24)
Statistical Analysis 1: Comparison: Inspiratory Muscle Training vs Control; Test type: Superiority; p = 0.005, Regression, Linear — p-value for MIP was adjusted by linear regression model
Statistical Analysis 2: Comparison: Inspiratory Muscle Training vs Control; Test type: Superiority; p = 0.038, Regression, Linear — adjusted p for MEP by linear regression

2. Secondary Outcome: Six Minutes Walking Distance
Description: The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes. The 6-minute walk distance (6 MWD) provides a measure for integrated global response of multiple cardiopulmonary and musculoskeletal systems involved in exercise.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: meter
Arm/Group | Control | Inspiratory Muscle Training
Number analyzed (Participants) | 13 | 13
meter
  baseline | 427 (125) | 411 (133)
  8 weeks | 447 (77) | 473 (117)
Statistical Analysis 1: Comparison: Control vs Inspiratory Muscle Training; Test type: Superiority; p = 0.063, Regression, Linear

3. Secondary Outcome: 6 Minute Work
Description: The 6-minute walk work (6Mwork) value was calculated as body mass distance covered during the 6-minute walking test.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Kg*Meter
Arm/Group | Control | Inspiratory Muscle Training
Number analyzed (Participants) | 13 | 13
Kg*Meter
  baseline | 20140 (7813) | 21052 (8286)
  8 weeks | 22457 (8596) | 23915 (8343)
Statistical Analysis 1: Comparison: Control vs Inspiratory Muscle Training; Test type: Superiority; p = 0.269, Regression, Linear

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Control | Inspiratory Muscle Training
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-31): https://cdn.clinicaltrials.gov/large-docs/18/NCT00952718/Prot_SAP_000.pdf